CLINICAL TRIAL: NCT05120284
Title: Trial of Dichloroacetate (DCA) in Glioblastoma Multiforme (GBM)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202101509; FD-R-007271-01 (Other Grant/Funding Number: Food and Drug Administration Research); PRO00034631 (Other: University of Florida-UFIRST); NCT05173623 (obsolete NCT alias)
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-03

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Dichloroacetic Acid; Genotype

STUDY DESIGN:
Intervention Model Description: subsequent ordered and alternating patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pre-Surgical Dichloroacetate (DCA) (Active Comparator): Study medication begins in subjects randomized to preoperative DCA. All subjects will be given the 12.5 mg/kg/12 hour DCA for pre-surgical dosing. Post-surgery the GSTZ1 haplotype will be utilized to dose all patients.
  Interventions: Drug: Dichloroacetate (DCA); Genetic: Genotype
- No Pre-Surgical Dichloroacetate (DCA) (Active Comparator): Subject randomized to start DCA after surgery will do so 12-24 hours postoperatively, depending on their ability to safely receive medication.
  Interventions: Drug: Dichloroacetate (DCA); Genetic: Genotype

INTERVENTIONS:
Drug: Dichloroacetate (DCA) — Study medication DCA is a liquid formulation mixed with an artificial sweetener containing aspartame and strawberry extract (50mg/mL)
  Participants will be genotyped to determine GSTZ1 (glutathione S-transferase Zeta-1) haplotype status, which will stratify this group into 1 of 2 dose regimens:
  EGT carriers will receive 12-14 mg/kg/12hr DCA. EGT non-carriers will receive 6-7 mg/kg/12 hr.
  Other Names: Sodium Dichloroacetate
Genetic: Genotype — Participants will be genotyped to determine GSTZ1 haplotype status.

SUMMARY:
Conduct a multicenter, open label Phase IIA trial of oral DCA in 40 surgical patients with recurrent GBM who have clinically indicated debulking surgery planned. No patients will be recruited at UF. Patients will be genotyped to establish safe dosing regimens and will be randomized to receive DCA (N=20) or no DCA (N=20) for one week prior to surgery. Deidentified blood and tumor tissue obtained at surgery will be assessed at UF for biochemical markers of DCA dynamics.

DETAILED DESCRIPTION:
Evaluate effects of dichloroacetate (DCA) on tumor PDC phosphorylation.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects will be male and female adults, aged 18 through 80 years, previously diagnosed with a GBM who have experienced tumor recurrence as determined by neuroimaging and some degree of symptomatology (e.g., headache, mental status change, seizure) and have clinically indicated tumor debulking surgery planned.
* All subjects will have completed initial, standard- therapy with surgical debulking, followed by radiation and temozolomide (TMZ) and will, therefore, be considered treatment failures. Patients with truly unmethylated GBM do not require prior treatment with temozolomide (TMZ).
* Patients will be recruited and studied at Johns Hopkins University, Johns Hopkins affiliated Sibley Memorial Hospital, and Wake Forest University. The DCA liquid formulation is on file with the FDA, is identical to that administered in our Phase I trial of brain tumor patients and can be given by mouth or feeding tube. Patients may retain whatever medications they are receiving for other conditions (e.g., hypertension, seizures), except patients requiring insulin or sulfonylurea therapy (see below).
* The probability of adverse drug-drug interactions is extremely low, for the following reasons. First, DCA is the only pharmaceutical in clinical use that is metabolized by GSTZ1. Second, DCA is not known to be metabolized by any other drug metabolizing enzyme system, thus precluding competition with other agents for biotransformation. Third, the results of both open label and randomized controlled trials of orally or parenterally administered DCA in the treatment of children and/or adults have never shown evidence of adverse drug-drug interactions (34). Thus, from decades of clinical investigations of use of DCA in various acutely or chronically ill populations, there is nothing to suggest adverse drug-drug interactions should be anticipated in this trial.
* Patients who are diabetic must have a screening hemoglobin A1c (Hgb A1c) level of at least 6.0.

Exclusion Criteria:

* Patients considered pre-terminal (life expectancy ≤ 2 months)
* Those who are pregnant will be excluded.
* DCA inhibits gluconeogenesis and lowers blood glucose levels in patients with type 2 diabetes. Therefore, in subjects who are receiving either insulin or a sulfonylurea, coadministration of DCA could lead to symptomatic hypoglycemia and those patients will be excluded from the trial.
* DCA is dialyzable and its clearance diminishes in patients with end stage renal failure (GFR ≤ 30 ml/min); such patients will be excluded from participating.
* DCA is metabolized by hepatic GSTZ1, so patients with severe liver insufficiency (total bilirubin > 2.0 mg/dl or ALT or AST > 3 x ULN) will be excluded.
* Patients with Hgb A1c level less than 6.0 at screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Level of phosphorylated PDC protein expressed in surgical tissue | Within 4 weeks post surgery
  The efficacy of dichloroacetate will be determined by the level of phosphorylated PDC protein expressed in surgical tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stacpoole, PhD, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Wake Forest University, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dunbar EM, Coats BS, Shroads AL, Langaee T, Lew A, Forder JR, Shuster JJ, Wagner DA, Stacpoole PW. Phase 1 trial of dichloroacetate (DCA) in adults with recurrent malignant brain tumors. Invest New Drugs. 2014 Jun;32(3):452-64. doi: 10.1007/s10637-013-0047-4. Epub 2013 Dec 3. PMID 24297161
- [Background] Patel MS, Korotchkina LG, Sidhu S. Interaction of E1 and E3 components with the core proteins of the human pyruvate dehydrogenase complex. J Mol Catal B Enzym. 2009 Nov 1;61(1-2):2-6. doi: 10.1016/j.molcatb.2009.05.001. PMID 20160912
- [Background] Stacpoole PW. The pyruvate dehydrogenase complex as a therapeutic target for age-related diseases. Aging Cell. 2012 Jun;11(3):371-7. doi: 10.1111/j.1474-9726.2012.00805.x. Epub 2012 Apr 4. PMID 22321732
- [Background] Kankotia S, Stacpoole PW. Dichloroacetate and cancer: new home for an orphan drug? Biochim Biophys Acta. 2014 Dec;1846(2):617-29. doi: 10.1016/j.bbcan.2014.08.005. Epub 2014 Aug 23. PMID 25157892
- [Background] DeBerardinis RJ, Chandel NS. Fundamentals of cancer metabolism. Sci Adv. 2016 May 27;2(5):e1600200. doi: 10.1126/sciadv.1600200. eCollection 2016 May. PMID 27386546
- [Background] Semenza GL. Oxygen sensing, homeostasis, and disease. N Engl J Med. 2011 Aug 11;365(6):537-47. doi: 10.1056/NEJMra1011165. No abstract available. PMID 21830968
- [Background] Brizel DM, Schroeder T, Scher RL, Walenta S, Clough RW, Dewhirst MW, Mueller-Klieser W. Elevated tumor lactate concentrations predict for an increased risk of metastases in head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2001 Oct 1;51(2):349-53. doi: 10.1016/s0360-3016(01)01630-3. PMID 11567808
- [Background] Walenta S, Wetterling M, Lehrke M, Schwickert G, Sundfor K, Rofstad EK, Mueller-Klieser W. High lactate levels predict likelihood of metastases, tumor recurrence, and restricted patient survival in human cervical cancers. Cancer Res. 2000 Feb 15;60(4):916-21. PMID 10706105
- [Background] Walenta S, Schroeder T, Mueller-Klieser W. Lactate in solid malignant tumors: potential basis of a metabolic classification in clinical oncology. Curr Med Chem. 2004 Aug;11(16):2195-204. doi: 10.2174/0929867043364711. PMID 15279558
- [Background] Park I, Larson PE, Zierhut ML, Hu S, Bok R, Ozawa T, Kurhanewicz J, Vigneron DB, Vandenberg SR, James CD, Nelson SJ. Hyperpolarized 13C magnetic resonance metabolic imaging: application to brain tumors. Neuro Oncol. 2010 Feb;12(2):133-44. doi: 10.1093/neuonc/nop043. Epub 2010 Jan 25. PMID 20150380
- [Background] Saraswathy S, Crawford FW, Lamborn KR, Pirzkall A, Chang S, Cha S, Nelson SJ. Evaluation of MR markers that predict survival in patients with newly diagnosed GBM prior to adjuvant therapy. J Neurooncol. 2009 Jan;91(1):69-81. doi: 10.1007/s11060-008-9685-3. Epub 2008 Sep 23. PMID 18810326
- [Background] Kahlon AS, Alexander M, Kahlon A, Wright J. Lactate levels with glioblastoma multiforme. Proc (Bayl Univ Med Cent). 2016 Jul;29(3):313-4. doi: 10.1080/08998280.2016.11929449. PMID 27365883
- [Background] Haas R, Cucchi D, Smith J, Pucino V, Macdougall CE, Mauro C. Intermediates of Metabolism: From Bystanders to Signalling Molecules. Trends Biochem Sci. 2016 May;41(5):460-471. doi: 10.1016/j.tibs.2016.02.003. Epub 2016 Feb 28. PMID 26935843
- [Background] Ippolito L, Morandi A, Giannoni E, Chiarugi P. Lactate: A Metabolic Driver in the Tumour Landscape. Trends Biochem Sci. 2019 Feb;44(2):153-166. doi: 10.1016/j.tibs.2018.10.011. Epub 2018 Nov 22. PMID 30473428
- [Background] Feron O. Pyruvate into lactate and back: from the Warburg effect to symbiotic energy fuel exchange in cancer cells. Radiother Oncol. 2009 Sep;92(3):329-33. doi: 10.1016/j.radonc.2009.06.025. Epub 2009 Jul 13. PMID 19604589
- [Background] Vegran F, Boidot R, Michiels C, Sonveaux P, Feron O. Lactate influx through the endothelial cell monocarboxylate transporter MCT1 supports an NF-kappaB/IL-8 pathway that drives tumor angiogenesis. Cancer Res. 2011 Apr 1;71(7):2550-60. doi: 10.1158/0008-5472.CAN-10-2828. Epub 2011 Feb 7. PMID 21300765
- [Background] Goodwin ML, Jin H, Straessler K, Smith-Fry K, Zhu JF, Monument MJ, Grossmann A, Randall RL, Capecchi MR, Jones KB. Modeling alveolar soft part sarcomagenesis in the mouse: a role for lactate in the tumor microenvironment. Cancer Cell. 2014 Dec 8;26(6):851-862. doi: 10.1016/j.ccell.2014.10.003. Epub 2014 Nov 26. PMID 25453902
- [Background] Sonveaux P, Vegran F, Schroeder T, Wergin MC, Verrax J, Rabbani ZN, De Saedeleer CJ, Kennedy KM, Diepart C, Jordan BF, Kelley MJ, Gallez B, Wahl ML, Feron O, Dewhirst MW. Targeting lactate-fueled respiration selectively kills hypoxic tumor cells in mice. J Clin Invest. 2008 Dec;118(12):3930-42. doi: 10.1172/JCI36843. Epub 2008 Nov 20. PMID 19033663
- [Background] Groussard C, Morel I, Chevanne M, Monnier M, Cillard J, Delamarche A. Free radical scavenging and antioxidant effects of lactate ion: an in vitro study. J Appl Physiol (1985). 2000 Jul;89(1):169-75. doi: 10.1152/jappl.2000.89.1.169. PMID 10904049
- [Background] Sattler UG, Mueller-Klieser W. The anti-oxidant capacity of tumour glycolysis. Int J Radiat Biol. 2009 Nov;85(11):963-71. doi: 10.3109/09553000903258889. PMID 19895273
- [Background] Calorini L, Peppicelli S, Bianchini F. Extracellular acidity as favouring factor of tumor progression and metastatic dissemination. Exp Oncol. 2012 Jul;34(2):79-84. PMID 23013757
- [Background] Gottfried E, Kunz-Schughart LA, Ebner S, Mueller-Klieser W, Hoves S, Andreesen R, Mackensen A, Kreutz M. Tumor-derived lactic acid modulates dendritic cell activation and antigen expression. Blood. 2006 Mar 1;107(5):2013-21. doi: 10.1182/blood-2005-05-1795. Epub 2005 Nov 8. PMID 16278308
- [Background] Goetze K, Walenta S, Ksiazkiewicz M, Kunz-Schughart LA, Mueller-Klieser W. Lactate enhances motility of tumor cells and inhibits monocyte migration and cytokine release. Int J Oncol. 2011 Aug;39(2):453-63. doi: 10.3892/ijo.2011.1055. Epub 2011 May 25. PMID 21617859
- [Background] Hirschhaeuser F, Sattler UG, Mueller-Klieser W. Lactate: a metabolic key player in cancer. Cancer Res. 2011 Nov 15;71(22):6921-5. doi: 10.1158/0008-5472.CAN-11-1457. PMID 22084445
- [Background] Vyas S, Zaganjor E, Haigis MC. Mitochondria and Cancer. Cell. 2016 Jul 28;166(3):555-566. doi: 10.1016/j.cell.2016.07.002. PMID 27471965
- [Background] Kaplon J, Zheng L, Meissl K, Chaneton B, Selivanov VA, Mackay G, van der Burg SH, Verdegaal EM, Cascante M, Shlomi T, Gottlieb E, Peeper DS. A key role for mitochondrial gatekeeper pyruvate dehydrogenase in oncogene-induced senescence. Nature. 2013 Jun 6;498(7452):109-12. doi: 10.1038/nature12154. Epub 2013 May 19. PMID 23685455
- [Background] Pate KT, Stringari C, Sprowl-Tanio S, Wang K, TeSlaa T, Hoverter NP, McQuade MM, Garner C, Digman MA, Teitell MA, Edwards RA, Gratton E, Waterman ML. Wnt signaling directs a metabolic program of glycolysis and angiogenesis in colon cancer. EMBO J. 2014 Jul 1;33(13):1454-73. doi: 10.15252/embj.201488598. Epub 2014 May 13. PMID 24825347
- [Background] Kamarajugadda S, Stemboroski L, Cai Q, Simpson NE, Nayak S, Tan M, Lu J. Glucose oxidation modulates anoikis and tumor metastasis. Mol Cell Biol. 2012 May;32(10):1893-907. doi: 10.1128/MCB.06248-11. Epub 2012 Mar 19. PMID 22431524
- [Background] Doherty JR, Cleveland JL. Targeting lactate metabolism for cancer therapeutics. J Clin Invest. 2013 Sep;123(9):3685-92. doi: 10.1172/JCI69741. Epub 2013 Sep 3. PMID 23999443
- [Background] Stacpoole PW. Therapeutic Targeting of the Pyruvate Dehydrogenase Complex/Pyruvate Dehydrogenase Kinase (PDC/PDK) Axis in Cancer. J Natl Cancer Inst. 2017 Nov 1;109(11). doi: 10.1093/jnci/djx071. PMID 29059435
- [Background] James MO, Jahn SC, Zhong G, Smeltz MG, Hu Z, Stacpoole PW. Therapeutic applications of dichloroacetate and the role of glutathione transferase zeta-1. Pharmacol Ther. 2017 Feb;170:166-180. doi: 10.1016/j.pharmthera.2016.10.018. Epub 2016 Oct 19. PMID 27771434
- [Background] Han Z, Berendzen K, Zhong L, Surolia I, Chouthai N, Zhao W, Maina N, Srivastava A, Stacpoole PW. A combined therapeutic approach for pyruvate dehydrogenase deficiency using self-complementary adeno-associated virus serotype-specific vectors and dichloroacetate. Mol Genet Metab. 2008 Apr;93(4):381-7. doi: 10.1016/j.ymgme.2007.10.131. Epub 2008 Feb 21. PMID 18206410
- [Background] Li J, Kato M, Chuang DT. Pivotal role of the C-terminal DW-motif in mediating inhibition of pyruvate dehydrogenase kinase 2 by dichloroacetate. J Biol Chem. 2009 Dec 4;284(49):34458-67. doi: 10.1074/jbc.M109.065557. Epub 2009 Oct 15. PMID 19833728
- [Background] Stacpoole PW. The dichloroacetate dilemma: environmental hazard versus therapeutic goldmine--both or neither? Environ Health Perspect. 2011 Feb;119(2):155-8. doi: 10.1289/ehp.1002554. Epub 2010 Oct 4. PMID 20920954
- [Background] Kaufmann P, Engelstad K, Wei Y, Jhung S, Sano MC, Shungu DC, Millar WS, Hong X, Gooch CL, Mao X, Pascual JM, Hirano M, Stacpoole PW, DiMauro S, De Vivo DC. Dichloroacetate causes toxic neuropathy in MELAS: a randomized, controlled clinical trial. Neurology. 2006 Feb 14;66(3):324-30. doi: 10.1212/01.wnl.0000196641.05913.27. PMID 16476929
- [Background] Shroads AL, Guo X, Dixit V, Liu HP, James MO, Stacpoole PW. Age-dependent kinetics and metabolism of dichloroacetate: possible relevance to toxicity. J Pharmacol Exp Ther. 2008 Mar;324(3):1163-71. doi: 10.1124/jpet.107.134593. Epub 2007 Dec 20. PMID 18096758
- [Background] Shroads AL, Langaee T, Coats BS, Kurtz TL, Bullock JR, Weithorn D, Gong Y, Wagner DA, Ostrov DA, Johnson JA, Stacpoole PW. Human polymorphisms in the glutathione transferase zeta 1/maleylacetoacetate isomerase gene influence the toxicokinetics of dichloroacetate. J Clin Pharmacol. 2012 Jun;52(6):837-49. doi: 10.1177/0091270011405664. Epub 2011 Jun 3. PMID 21642471
- [Background] Abdelmalak M, Lew A, Ramezani R, Shroads AL, Coats BS, Langaee T, Shankar MN, Neiberger RE, Subramony SH, Stacpoole PW. Long-term safety of dichloroacetate in congenital lactic acidosis. Mol Genet Metab. 2013 Jun;109(2):139-43. doi: 10.1016/j.ymgme.2013.03.019. Epub 2013 Apr 6. PMID 23611579
- [Background] Vallee A, Guillevin R, Vallee JN. Vasculogenesis and angiogenesis initiation under normoxic conditions through Wnt/beta-catenin pathway in gliomas. Rev Neurosci. 2018 Jan 26;29(1):71-91. doi: 10.1515/revneuro-2017-0032. PMID 28822229
- [Background] Velpula KK, Guda MR, Sahu K, Tuszynski J, Asuthkar S, Bach SE, Lathia JD, Tsung AJ. Metabolic targeting of EGFRvIII/PDK1 axis in temozolomide resistant glioblastoma. Oncotarget. 2017 May 30;8(22):35639-35655. doi: 10.18632/oncotarget.16767. PMID 28410193
- [Background] Schwartz L, Seyfried T, Alfarouk KO, Da Veiga Moreira J, Fais S. Out of Warburg effect: An effective cancer treatment targeting the tumor specific metabolism and dysregulated pH. Semin Cancer Biol. 2017 Apr;43:134-138. doi: 10.1016/j.semcancer.2017.01.005. Epub 2017 Jan 22. PMID 28122260
- [Background] Rubinstein LV, Steinberg SM, Kummar S, Kinders R, Parchment RE, Murgo AJ, Tomaszewski JE, Doroshow JH. The statistics of phase 0 trials. Stat Med. 2010 May 10;29(10):1072-6. doi: 10.1002/sim.3840. PMID 20419759